CLINICAL TRIAL: NCT05936424
Title: Investigating the Effects of Menstrual Cycle Phase Based Training on Muscle Strength and Hypertrophy
Brief Title: Menstrual Cycle Phase Based Training
Acronym: MCPBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Stuart Phillips, Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 16355
Record Dates: First submitted 2023-06-22; First posted 2023-07-07 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Menstrual Cycle; Resistance Exercise

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial (RCT), within-between subject design. Legs will be randomized to one of four groups: non-exercise control (CON), exercise control (EX), Follicular based training (FOL), Luteal based training (LUT)
Masking Description: As this is a resistance exercise training intervention, participants will be unable to be masked to their treatment condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Non-Exercise Control (CON) (Active Comparator): This condition will serve as a non-exercise control and will not be performing resistance exercise training (RET)
  Interventions: Other: Non-Exercise Control Leg
- Follicular Based Training (FOL) (Experimental): This condition will have high volume of RET (20 weekly sets) during the follicular phase and low volume during the luteal phase of the participant's menstrual cycle.
  Interventions: Other: Unilateral Resistance Exercise Leg
- Luteal Based Training (LUT) (Experimental): This condition will have high volume of RET (20 weekly sets) during the luteal phase and low volume during the follicular phase of the participant's menstrual cycle.
  Interventions: Other: Unilateral Resistance Exercise Leg
- Exercise Control (EX) (Experimental): This condition will have consistent training volume (12 weekly sets) throughout the duration of the study, regardless of what phase of the menstrual cycle the participant is in.
  Interventions: Other: Unilateral Resistance Exercise Leg

INTERVENTIONS:
Other: Unilateral Resistance Exercise Leg — One will perform unilateral resistance exercise
  Arms: Exercise Control (EX); Follicular Based Training (FOL); Luteal Based Training (LUT)
Other: Non-Exercise Control Leg — One leg will serve as a non-exercise control
  Arms: Non-Exercise Control (CON)

SUMMARY:
The primary purpose of this study is to employ state-of-the-art methods to fill current knowledge gaps on the effects of the menstrual cycle on resistance exercise training adaptations. This work will reduce the sex gap present in exercise physiology, improving women's health information by yielding a deeper understanding of the effect of female physiology on exercise adaptations and subsequent health benefits.

Employing a unilateral training design, participant's will have their legs randomized to one of four groups: non-exercise control (CON), exercise control (EX), Follicular based training (FOL), Luteal based training (LUT)

Researchers will compare these conditions to see if there are greater benefits to prioritizing resistance training around phases of the menstrual cycle,

DETAILED DESCRIPTION:
Participants will be required to track their menstrual cycle (MC) for a total of four MC's. MC tracking will be done via self-reported menstrual onset and ovulation strips. During the first tracking cycle participants will be asked to come in at three time points for blood draws to confirm hormone concentrations and familiarize them with the strength testing protocol. Following the tracking month participant legs will then be blocked randomized based on leg skeletal muscle mass and strength into one of four groups: non-exercise control (CON), exercise control (EX), follicular based training (FOL) and luteal based training (LUT). Participants will then be asked to come in ~2x per week (4-6x/menstrual cycle phase) for resistance training under direct supervision. Participants will be trained in unilateral leg extension and unilateral leg press. For legs randomized to the FOL and LUT group, training volume will be manipulated by changing the number of sets completed. The FOL group will train high volume (~20+ sets per week) in their follicular phase and low volume (~5 sets/week) in their luteal phase, the opposite will be true for the LUT group. Muscle biopsies will be taken both prior to and after training to assess changes in fiber cross-sectional area (CSA) and capillarization. Segmental body composition will be assessed both prior and post training using bioelectrical impedance analysis (BIA), dual x-ray absorptiometry (DXA), and vastus lateralis cross-sectional area and thickness. Muscle strength will also be assessed pre and post training using the isokinetic dynamometer, unilateral one-repetition maximum (1RM) leg extension and unilateral 1RM leg press.

ELIGIBILITY:
Inclusion Criteria:

* Women, between the ages of 18 - 30 years (inclusive)
* Have a body mass index (BMI) between 18-35 kg·m2 (inclusive)
* Be in general good health as assessed by a general health questionnaire
* Non-smoking
* Regular menstrual cycle (21-35 days, inclusive)
* Not using hormonal contraceptives
* Willing and able to provide informed consent

Exclusion Criteria:

* Use of tobacco or related products.
* Ineligible to participate in physical activity based on get active questionnaire (GAQ)
* Any concurrent medical, orthopedic, or psychiatric condition that, in the opinion of the Investigator, would compromise his/her ability to comply with the study requirements.
* Current illnesses which could interfere with the study (e.g. prolonged severe diarrhea, regurgitation, difficulty swallowing)
* Use of hormonal contraceptives
* Currently pregnant
* Training more than 3x/week for the past 6 months.
* Have any electronic medical or metal implants
* A history of neuromuscular disorders or muscle/bone wasting diseases
* The use of any medications known to affect protein metabolism (glucocorticoids, non-steroidal anti-inflammatory medication, or prescription strength acne medication, etc.)
* A (family) history of thrombosis
* The use of anticoagulant medications
* Excessive alcohol consumption (>21 units/wk)
* History of bleeding diathesis, platelet or coagulation disorders, or antiplatelet/anticoagulation therapy

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Muscle Hypertrophy | 16 weeks
  The investigators will be measuring participant's muscle cross-sectional area of the quadriceps pre and post training intervention via ultrasound (US)
  US is used to measure skeletal muscle thickness and cross-sectional area. A trained and experienced study investigator will perform the US measures. US will be used to measure the cross-sectional area of the vastus lateralis muscle on both legs. After remaining supine for 15-minute, your feet will be positioned in a custom foot-hold apparatus that prevents depression of the thigh against the bed. Mid-thigh will be identified via palpation. A marker will be used to draw a line down your leg, perpendicular to the surface of the bed, and horizontal markings will be made every 2 cm serving as a guideline for ultrasound probe placement. Ultrasound images will be taken at each horizontal marking and used to measure the muscle cross-sectional area of the quadriceps.
Muscular Strength | 16 Weeks
  The investigators will be measuring participant's muscle strength via one-repetition maximum testing using the unilateral leg press.

CONTACTS AND LOCATIONS:
Locations (1):
- Exercise Metabolism Research Laboratory, McMaster Univeristy, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
All participants will be assigned a unique subject identification number (ID), and therefore, other researchers involved with analyses will not have access to identifying participant information.